CLINICAL TRIAL: NCT05846126
Title: Digital Rehabilitation With Cognitive Training, Physical Activity and Mindfulness for People With Post-acute COVID-19 Syndrome With Cognitive Impairment. REHABCOVID Project.
Brief Title: Digital Multimodal Rehabilitation for People With Post-acute COVID-19 Syndrome.
Acronym: REHABCOVID
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Consorci Sanitari de Terrassa (Other)
Collaborators: University of Barcelona (Other); Universitat de Girona (Other); Unitat Assistencial i Preventiva de l'Esport- Centre d'Alt rendiment (Unknown); Universitat Politècnica de Catalunya (Other); Corporación Fisiogestión (Unknown)
Responsible Party: Principal Investigator, Maite Garolera, Principal Investigator of the Brain, Cognition, and Behavior Research Group (C3-CST)., Consorci Sanitari de Terrassa
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: TED2021-130409B-C51
Record Dates: First submitted 2023-05-04; First posted 2023-05-06 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Post-COVID Syndrome
Keywords: COVID-19; Immersive Virtual Reality; Cognition; Cognitive Training; Physical Exercise; Mindfulness
MeSH Terms: conditions — COVID-19; Motor Activity

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Telematic group (Experimental): This program combines cognitive training, physical exercise, and mindfulness tasks delivered remotely to participants. The cognitive training includes 24 interactive sessions over 12 weeks aimed at training attention, memory, and executive function. The physical exercise program is personalized and includes balance work, stretching, and muscle strengthening exercises, with two sessions per week for 12 weeks. The mindfulness component adapts the Mindfulness-Based Stress Reduction program, including body scanning, seated meditation, and gentle Hatha yoga, with one supervised session per week via video call over 12 weeks. The program is designed for autonomous use by participants.
  Interventions: Behavioral: RehabCovid_Telematic
- Immersive Virtual Reality group (Experimental): The sessions will consist of carrying out a face-to-face multimodal stimulation program with the application of MK360 immersive technology for the cognitive, emotional, behavioral, physical, functional - social areas. The multimodal intervention includes 24 interactive sessions two sessions per week, over 12 weeks. They will follow the following scheme:
  1. Welcome and awareness of the here and now.
  2. Physical activation.
  3. Cognitive stimulation.
  4. Relaxation techniques and Mindfulness.
  5. Feedback and end of session.
  During the intervention period, patients will be provided with a downloadable App with a username and password, so they can access it. From the App, they will view the tests to answer according to tempos and therapeutic direction.
  Interventions: Behavioral: RehabCovid_ImmersiveVR
- Active control program (Active Comparator): In paper or pdf format, patients in the active control group will receive guidelines for physical and cognitive stimulation to do autonomously at home. Patients in the active control group will receive guidelines for cognitive and physical stimulation and meditation exercises in paper or pdf format, to be done independently at home. They will be encouraged to do physical exercises, meditation, and cognitive activities two times a week.
  Interventions: Behavioral: Control_Condition

INTERVENTIONS:
Behavioral: RehabCovid_Telematic — A multimodal and digitally-based cognitive training, physical exercise, and mindfulness intervention delivered remotely.
  Arms: Telematic group
Behavioral: RehabCovid_ImmersiveVR — A multimodal and digitally-based cognitive training, physical exercise and mindfulness intervention delivered face to face and through 360MK Virtual Reality technology
  Arms: Immersive Virtual Reality group
Behavioral: Control_Condition — Traditional paper or pdf format multimodal intervention that will combine cognitive, mediation and physical activities.
  Arms: Active control program

SUMMARY:
Although most infected people survive the infection, many have persistent sequelae or symptoms, which cause disability or decreased quality of life. The World Health Organization has called on countries to prioritize the rehabilitation of the consequences of COVID-19 in both the medium and long term, as this chronicity is expected to impact the health public and the economy in the coming years.

RehabCOVID (also referred to as RehabNautilus) is born from the need to provide solutions to persistent cognitive impairment symptoms of people who have suffered from COVID-19. Thus, we will offer people with long COVID that accomplish inclusion/exclusion criteria to participate in a randomized clinical trial to evaluate the effectiveness of cognitive stimulation therapy combined with physical exercise and mindfulness. The current project is a single-blind randomized control study, where we will compare two combined interventions with a control group that will encompass different functional, structural, and biochemical changes and interactions in the brain. We will study the effects that this combined intervention produces in the brain. We expect to gain more insight into the specific neuroplasticity mechanisms of cognitive persistent COVID symptoms.

DETAILED DESCRIPTION:
The current project is a single-blind randomized clinical study, where we will compare two combined interventions with a control group that will encompass different functional, structural, and biochemical changes and interactions in the brain. We will study the effects that this combined intervention produces in the brain. We expect to gain more insight into the specific neuroplasticity mechanisms of cognitive persistent COVID symptoms.

Specifically, we aim to:

1. Examine the effects of a combined intervention in a population of long-COVID patients on various domains: cognition; emotion; physical health and quality of life.
2. Study the molecular mechanisms (biomarkers of inflammation, vascular risk, growth factors, angiogenesis, neurogenesis, and cellular metabolism markers of neural plasticity) by which the combined interventions influence brain functions.
3. Compare the levels of neural plasticity-related miRNAs and Sirt-1 protein in the plasma of long-COVID patients of the experimental groups versus the active control group.
4. Examine specific plasticity effects of each of the two interventions regarding structural magnetic resonance imaging (MRI) combined with volumetry and morphometry, resting-state functional MRI.
5. Determine the influence that demographic characteristics, previous pathologies, lifestyle, baseline brain state, and genetic polymorphisms can have on neuroplasticity.

We hypothesize that we will find recovery in our three groups, although it will be enhanced in the two experimental groups (those that combine cognitive training with physical activity and mindfulness) compared to our control group.

1. Post-COVID patients of the experimental groups will perform better than those patients of the active control group in cognition (episodic memory tests, executive function, attention, and speed processing), functional capacity, mental health, and quality of life measures at the end of the intervention.
2. Post-COVID patients of the experimental groups will show greater changes in biomarkers than those patients of the active control group at the end of the intervention. These changes will include higher levels of Sirt-1 and regulation of neural plasticity-related miRNAs in plasma from patients in the experimental group.
3. We will find an association between changes in biomarkers and cognitive, functional capacity and mental health outcomes in individuals of the experimental groups.
4. Post-COVID patients of the experimental groups will show greater improvements in grey and white matter structural data and functional connectivity than those patients of the active control group at the end of the intervention.

ELIGIBILITY:
Inclusion Criteria:

* Over 18 years old.
* Participants with a diagnosis of COVID-19 presenting persistent neurological symptoms at least 12 weeks after acute infection.
* They will have cognitive complaints
* Consent from a physician to engage in an exercise intervention

Exclusion Criteria:

* Established diagnosis before COVID-19 disease of psychiatric, neurological, developmental disorder, or systemic pathologies are known to cause cognitive deficits.
* Motor or sensory alterations that impede the rehabilitation program.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 158 (Estimated)
Dates: Start 2023-05-01 (Actual); Primary Completion 2024-09-30 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Differences between groups in scores of global cognition | Before the intervention and 12 weeks later
  Global cognition was assessed with the Montreal Cognitive Assessment (MoCA) a screening tool designed to identify mild cognitive impairment (MCI) and other cognitive deficits. The MoCA takes around 10-15 minutes to complete and consists of 30 items (range=0-30). Higher scores mean a better outcome.
Differences between groups in scores of selective attention, inhibition, and processing speed | Before the intervention and 12 weeks later
  Selective attention, inhibition, and processing speed are measured with the Stroop Color and Word Test. Participants are asked to name the color of a series of color patches (Stroop Color Naming), read a series of color words (Stroop Word Reading), and name the color of a series of color words where the word and color do not match (e.g., the word "red" written in blue ink), Stroop Color-Word Interference. Higher scores mean a better outcome.
Differences between groups in scores of Visual scanning and processing speed | Before the intervention and 12 weeks later
  Visual scanning and processing speed are measured with the Trail-Making Test-A version. Participants are asked to connect a series of numbered circles on a page in numerical order. Higher scores mean a better outcome.
Differences between groups in scores of Executive functioning and cognitive flexibility | Before the intervention and 12 weeks later
  Executive functioning and cognitive flexibility are measured with the Trail-Making Test-B version. Participants are asked to connect a series of circles that contain both numbers and letters in alternating numerical and alphabetical order. Higher scores mean a better outcome.
Differences between groups in scores of auditory attention | Before the intervention and 12 weeks later
  Auditory attention is measured with Digit Span Forward from WAIS-IV. Participants are asked to repeat numbers in the same order as read aloud by the examiner. Higher scores mean a better outcome.
Differences between groups in scores of working memory_DSB | Before the intervention and 12 weeks later
  Working memory is measured with Digit Span Backward from WAIS-IV. Participants are asked to repeat the numbers in the reverse order of that presented by the examiner. Higher scores mean a better outcome.
Differences between groups in scores of Perceptual Reasoning | Before the intervention and 12 weeks later
  Perceptual Reasoning is measured with Matrices from the WAIS-IV. Participants are presented with a pattern or design with one missing piece and are asked to select the correct piece from a set of options to complete the pattern. Higher scores on the Perceptual Reasoning Index mean a better outcome.
Differences between groups in scores of sustained attention and impulsivity | Before the intervention and 12 weeks later
  Conners Continuous Performance Test - 2nd edition (CPT-II) is task-oriented computerised assessment of attention-related problems. Participants are presented with a repetitive array of visual stimuli on a computer screen for 14 min. Participants are instructed to press the space bar every time a letter other than "X" appears and to not press the space bar when "X" appears. The rate of stimulus presentation varies according to 1, 2, and 4 s intervals throughout the task. Measures: Correct Detection (Higher rates indicate better outcome), Reaction times (Lower scores indicate better outcome), Omission errors (Lower rates indicate better outcome), and Commission errors (Lower rates indicate better outcome).
Differences between groups in scores of processing speed | Before the intervention and 12 weeks later
  The Digit Symbol Coding subtest from the WAIS-III is a neuropsychological assessment instrument for the detection of brain dysfunction in children and adults. It consists of replacing symbols that lack verbal meaning with numbers based on a key. Higher scores indicate better outcomes.
Differences between groups in scores of verbal memory and learning | Before the intervention and 12 weeks later
  Verbal memory and learning are measured with the Rey Auditory Verbal Learning Test (RAVLT). It is a word-learning test where five presentations of a 15-word list are given, each followed by an attempted recall. This is followed by a second 15-word interference list (list B), followed by a recall of list A. Delayed recall and recognition are also tested. Higher scores mean a better outcome.
Differences between groups in scores of phonetic fluency | Before the intervention and 12 weeks later
  Phonetic fluency is measured with the FAS test. It consists of saying words that start with a certain letter, as many words as possible must be mentioned during a specific time of 1 minute. The standard administration of the test provides three letters, the most used are the letters F, A, and S. Higher scores indicate better performance.
Differences between groups in scores of semantic verbal fluency | Before the intervention and 12 weeks later
  Semantic verbal fluency is measured with the ANIMAL test. It consists of generating the name of as many species of animals as possible within 1min. Higher scores indicate better performance.
Differences between groups in scores of memory and everyday forgetfulness | Before the intervention and 12 weeks later
  Memory and everyday forgetfulness are measured with The Memory Failures of Everyday-MFE Questionnaire is a self-reported test that allows an assessment of memory and everyday forgetfulness. It is a unifactorial questionnaire and consists of 30 items. The total score results from the sum of the scores in each item, from 1 to 30. The MFE can assess the current situation of the patients and their evolution long-term or changes due to treatment. Scores <8 represent an optimal memory function. Lower scores indicate better outcomes.

SECONDARY OUTCOMES:
Differences between groups in scores of anxiety | Before the intervention and 12 weeks later
  Anxiety is measured with the 7-item Generalized Anxiety Disorder Scale (GAD-7), a Likert-type scale with questions ranging from "not at all" (0 points) to "nearly every day" (3 points). The maximum score is 24. Higher scores mean a worse outcome.
Differences between groups in scores of depression | Before the intervention and 12 weeks later
  Depression is measured with the Patient Health Questionnaire-9 (PHQ-9) which scores each of the 9 DSM-IV criteria as "not at all" (0 points) to "nearly every day" (3 points). Higher scores mean a worse outcome.
Differences between groups in scores of Mindfulness levels | Before the intervention and 12 weeks later
  Mindfulness levels are measured with The Mindful Attention Awareness Scale (MAAS) assesses an individual's level of mindfulness, including attention, awareness, and non-judgment. The 15-item self-report questionnaire uses a 6-point Likert scale to measure an individual's general tendency to be aware of and attentive to their current experience. Scores on the MAAS range from 15 to 90, with higher scores indicating greater levels of mindfulness. A higher score suggests better outcome.
Differences between groups in scores of Fatigue | Before the intervention and 12 weeks later
  Fatigue is measured with the Chalder Fatigue Scale, an 11-item questionnaire measuring the severity of physical and mental fatigue on two separate subscales. Seven items represent physical fatigue (items 1-7) and 4 represent mental fatigue (items 8-11). Each item " less than usual" (0) to " much more than usual" (3). The ratings of items are added together to calculate the total score (range=0-33). High scores represent high levels of fatigue.
Differences between groups in scores of psychological flexibility | Before the intervention and 12 weeks later
  Psychological flexibility is measured with the Acceptance and Action Questionnaire, a 7-point Likert scale, ranging from 1 ("never true") to 7 ("always true"), indicating how frequently they experience the described behavior or feeling in their daily lives. The scale has 9 items and the total score ranges from 9 to 63, with higher scores indicating greater levels of psychological flexibility (better outcome).
Differences between groups in Functionality | Before the intervention and 12 weeks later
  Functionality is measured with a 12-item World Health Organization Disability Assessment Schedule-II (WHODAS-II). Patients are asked to state the level of difficulty experienced, considering how they usually do the activity. The scale scores each item as "none" (1) to "cannot do" (5). The total score is calculated with an SPSS syntax, and the range varies from 0 to 100, with higher scores reflecting more significant disability.
Differences between groups in scores of Sleep Quality | Before the intervention and 12 weeks later
  Sleep Quality is measured with The Pittsburgh Sleep Quality Index (PSQI). This test presents 24 items, although only 19 are taken into account for the correction. This test is divided into 7 dimensions, namely, sleep quality, sleep onset latency, sleep duration, sleep efficiency, sleep disturbances, hypnotic drugs, and daytime dysfunction. Higher scores indicate worse sleep quality.
Differences between groups in scores of Quality of Life | Before the intervention and 12 weeks later
  Quality of Life is measured with EuroQol a self-completion questionnaire, which consists of five questions: covering mobility, hygiene, activities, pain, and anxiety. The descriptive system divides each of the 5 dimensions into three levels of response: the absence of a problem, some problem, and extreme problem. Lower scores indicate better outcomes. In addition, the questionnaire has a plus scale where the participants rated their health state on a scale of 0-100. In this scale, higher scores indicate better outcome.
Differences between groups in scores of performed physical activity | Before the intervention and 12 weeks later
  Performed physical activity is measured with The International Physical Activity Questionnaire (IPAQ) is a questionnaire composed of 7 questionsin order to assessthe frequency, duration, and intensity (vigorous or moderate) of the performed physical activity, walking, and sitting time during a business day for the last 7 days. Later, from the minutes obtained from the participant's answers, the METS (metabolic equivalent tasks) conversion is performed, allowing a classification, depending on the energy consumption obtained for each activity, into three categories (low, medium, high). Higher score indicate better outcome.
Differences between groups in White Matter integrity | Before the intervention and 12 weeks later
  White matter integrity: tractography measured by MRI
Differences between groups in brain Volumetry | Before the intervention and 12 weeks later
  Grey and white matter volume measured by MRI
Differences between groups in Resting-state connectivity | Before the intervention and 12 weeks later
  Resting state brain activity using fMRI
Differences between groups in rate of expression analysis of Sirt-1 levels | Before the intervention and 12 weeks later
  Sirt-1 levels are measured with the Sirtuin-1 ELISA Kit
Differences between groups in rate of expression analysis of different microRNAs | Before the intervention and 12 weeks later
  microRNAs are measured with TaqMan miRNA qRT-PCR

CONTACTS AND LOCATIONS:
Locations (1):
- Consorci Sanitari de Terrassa, Terrassa, Spain

IPD SHARING:
Plan to Share IPD: No